CLINICAL TRIAL: NCT00893750
Title: Effects of Trauma-Therapy and Truth Education, Conflict Resolution and Social Skills Trainings and Traditional Ways of Coping in Northern Uganda
Brief Title: Trauma and Truth Interventions (NET) Versus Conflict Resolution and Social Skills Trainings for Vulnerable Youths in Northern Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Prof. Dr. Thomas Elbert, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NE1390/2.1_UKon
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: PTSD; Depression; Aggression
Keywords: Vulnerable Youths in Northern Uganda; Formerly Abducted Children; Reintegration and Reconciliation; Trauma Treatment; Narrative Exposure Therapy; Reconciliation; Revenge Feelings
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NET Truth Education (Experimental)
  Interventions: Behavioral: NET Truth Education
- Conflict Resolution Trainings (Experimental)
  Interventions: Behavioral: Conflict Resolution and Social Competence Skills
- Traditional Methods (Experimental)
  Interventions: Behavioral: Traditional Ways of Coping

INTERVENTIONS:
Behavioral: NET Truth Education — Individual Narrative Exposure and Truth Education in Groups
  Arms: NET Truth Education
Behavioral: Conflict Resolution and Social Competence Skills — Conflict Resolution and Social Competence Skills in Groups
  Arms: Conflict Resolution Trainings
Behavioral: Traditional Ways of Coping — Methods Collected by Local Teachers to Help Vulnerable Children and Youths in Northern Uganda
  Arms: Traditional Methods

SUMMARY:
More than 300,000 children are fighting in armed conflicts all over the world. In Uganda an estimated number of 25,000 children have been abducted and forced to fight or work as porters and sex slaves on the side of the rebels during the conflict between the Lord's Resistance Army (LRA) and the Ugandan government. Each year, thousands of former child soldiers have returned to their communities after they had fled or were freed from the rebels. It is well known that a high percentage of these youths are suffering from mental health problems. This could be one of the possible reasons why they are facing difficulties to reintegrate into their communities.

The main aim of the proposed project is two-fold. On the one hand, the investigators want to systematically explore the relationship between mental health and important variables for reintegration into the communities like aggression, hostility, feelings of revenge, compromises and conflict behaviour and readiness for reconciliation in formerly abducted and other vulnerable youth (orphans, child mothers and handicapped youths) in Northern Uganda. On the other hand, the investigators want to probe the efficacy of existing and newly developed interventions for formerly abducted and other vulnerable youths that are supposed to foster their mental well-being as well as their reintegration into the society and therewith are part of the long-term prevention of new conflicts in Northern Uganda.

ELIGIBILITY:
Inclusion Criteria:

* for individual NET Treatment: PTSD diagnosis
* for group interventions: all youths in the selected vocational training centres will be included

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms and Functional Level | 6-months and 12-months follow-up

SECONDARY OUTCOMES:
Aggression Reconciliation Re-Integration Conflict and Compromise Behaviour | 6-months and 12-months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Vivo, Gulu & Kitgum, Uganda

REFERENCES:
- See also: NGO — http://www.vivo.org